CLINICAL TRIAL: NCT01164397
Title: Efficiency of Rosuvastatin Versus the Fixed Combination of Ezetimibe/Simvastatin to Reduce the Cholesterol Levels in Outpatients in a Realistic Environment. A Retrospective Study
Brief Title: Efficiency of Rosuvastatin Versus the Fixed Combination of Ezetimibe/Simvastatin in Outpatients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CME-CRE-2010/1; DM-CRESTOR-0003 (Other: AstraZeneca)
Record Dates: First submitted 2010-05-28; First posted 2010-07-16 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Dyslipidemia
Keywords: Hypercholesterolemia; Statins
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dislipidemic Population: People with high levels of total cholesterol, LDL, C-HDL and triglycerides

SUMMARY:
The aim of this study is to evaluate the effectiveness of Rosuvastatin versus Ezetimibe/Simvastatin in dyslipidemic patients treated for at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Dislipidemic population treated with rosuvastatin or ezetimibe/simvastatin for at least for 8 weeks
* Who have completed at least 80% of the treatment
* To have determinations at least of CT, TG C-LDL and CHDL before starting treatment and after 8 weeks of taking the medicine

Exclusion Criteria:

* Initiating different therapy lipid lowering to Rosuvastatin or Ezetimibe/Simvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Care clinic private practice
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2009-04; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The percentage of the patients that achieve the goal proposed for NCEP ATP III (2001 y 2004) will be assessed, to C-LDL in patients treated with Rosuvastatin or Ezetimibe/Simvastatin at least for 8 weeks. | Data will be collected using CRFs after complete at least 15 patients over a 24 week period.

SECONDARY OUTCOMES:
The percentage of LDL-C reduction according to baseline levels in patients treated wuth Rosuvastatin or Ezetimibe/Simvastatin for at least 8 weeks. | Data will be collected using CRFs after complete at least 15 patients over a 24 week period.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Polanco, MD, Study Director — AstraZeneca
Locations (9):
- Mexico (9):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Cuernavaca, Morelos
  - Research Site, Monterrey, Nuevo León
  - Research Site, Puebla City, Puebla
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Veracruz, Xalapa
  - Research Site, Mérida, Yucatán
  - Research Site, Durango